CLINICAL TRIAL: NCT01139177
Title: SAMBA EU Femoropopliteal Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NovoStent Corporation (Industry)
Responsible Party: Earle Canty, VP RACAQA, NovoStent Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60-00857-01
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Peripheral Vascular Disease
Keywords: Peripheral vascular disease - SFA and popliteal arteries.
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stent placement (Experimental)
  Interventions: Device: Stenting of atherosclerotic lesion(s)

INTERVENTIONS:
Device: Stenting of atherosclerotic lesion(s) — Stenting of atherosclerotic lesions post pre-dilatation of lesion(s)
  Other Names: SAMBA Stent and Delivery System

SUMMARY:
The primary objective of this study is to evaluate the safety and performance of the SAMBA Stent and Delivery System in the treatment of femoropopliteal lesions.

ELIGIBILITY:
Inclusion Criteria:

Screening

1. Patient must be ≥ 21 years of age with life expectancy > 1 year.
2. Symptomatic leg ischemia requiring treatment of the superficial femoral and/or popliteal artery (Rutherford category 2-4; claudication, rest pain).
3. Patient must be a suitable candidate for PTA and stenting.
4. Patient is willing and able to return to the site of the investigation at the specified study intervals and undergo follow-up requirements.
5. The patient or legal representative has provided written informed consent using a form that is reviewed and approved by the EC for the Clinical Site.

Pre-Intervention

1. Target lesion has ≥ 50% stenosis as demonstrated angiographically.
2. Lesion length ≤ 15 cm.
3. Reference vessel diameter of 5 to 6 mm.
4. Patient has at least 1 vessel run-off prior to treatment.

Exclusion Criteria:

Screening

1. The subject is pregnant or will become pregnant during the study or has any other condition that would preclude having x-rays. (Pre-menopausal women must have a negative pregnancy test within 7 days of the procedure.)
2. Patients who have experienced a cardiovascular accident (CVA) or a myocardial infarction (MI) within 3 months prior to the procedure.
3. Subject has had or plans to have a surgical or interventional procedure within 30 days before or after the implantation procedure of the SAMBA Stent.
4. Existing hemorrhagic disease or coagulation problems or inability to take dual anti-platelet therapy.
5. Contrast allergy that cannot be corrected with medication (e.g. steroids, etc.).
6. Subject has other medical, social, or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment and the procedures and evaluations pre- and post-treatment.
7. Patient is currently participating in another investigational drug or device study.

Pre-Intervention

1. Uncorrectable severe aorto-iliac occlusive disease or severe common femoral artery stenosis preventing access or limiting inflow (e.g., stenosis greater than 50%).
2. Uncorrectable occlusive disease limiting outflow (e.g., stenosis greater than 50%)
3. Patients with previous surgery in the target vessel or stent that will be closer than 2 cm to either edge of SAMBA Stent(s).
4. Lack of 1 cm of healthy vessel proximal to proximal target
5. Lack of popliteal reconstitution (at least 2 cm of normal distal popliteal).
6. Inability to cross the lesion with a guidewire.
7. More than 1 lesion in the same limb requiring treatment that will not be covered by continuous stenting.
8. Unsuccessful balloon pre-dilation (i.e., the residual stenosis is greater than 30%).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is defined as freedom from all cause death, unplanned index limb amputation, and target lesion revascularization. | through 30 days
The primary efficacy endpoint is defined as stent patency via Color Duplex Ultrasound (Peak Velocity Ratio ≤ 2.5). | 3 months

SECONDARY OUTCOMES:
Clinically-Driven Target Lesion Revascularization (i.e., with documented preintervention evidence of at least 50% diameter stenosis (quantitative angiographic ≥ 50% or PSVR > 2.5). | 12 months
Change in Rutherford Classification compared to pre-implant. | 12 months
Stent Patency via Color Duplex Ultrasound (Peak Systolic Velocity Ratio ≤ 2.5). | 12 months
Stent Fractures. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Herz-Zentrum Leipzig
Locations (2):
- Germany (2):
  - Herz Zentrum Bad Krozingen, Bad Krozingen
  - Herz-Zentrum Leipzig, Leipzig